CLINICAL TRIAL: NCT05958173
Title: Biomechanical, Neurophysiological and Clinical Effects of 6-month Stimulation Using TRPV1 and TRPA1 Agonists in Older Patients With Oropharyngeal Dysphagia
Brief Title: Effects of 6-month of Treatment With TRPV1 and TRPA1 Agonists in Older Patients With OD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, Principal Investigator, Hospital de Mataró
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI22/01101
Record Dates: First submitted 2023-05-23; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Oropharyngeal Dysphagia; Swallowing Disorder
Keywords: TRP agonists; Sensory stimulation; Rehabilitation
MeSH Terms: conditions — Deglutition Disorders | interventions — Capsaicin; piperine

STUDY DESIGN:
Intervention Model Description: Single-center, double-blinded, three-arm randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: The products will be prepared in the Pharmacy Department and will be labeled with a code that does not allow its identification neither by the patient nor by the investigator who administers it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Capsaicin (Active Comparator): Natural TRPV1 agonist at a concentration of 10mcM. Posology: 10 mL every 8h for 6 month.
  Interventions: Dietary Supplement: Capsaicin
- Piperine (Active Comparator): Natural TRPA1/V1 agonist at a concentration of 150mcM. Posology: 10 mL every 8h for 6 month.
  Interventions: Dietary Supplement: Piperine
- Placebo (Placebo Comparator): Deionized water + the same preservatives as in the active treatments
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Capsaicin — Oral stimulation with natural TRPV1 agonist
  Arms: Capsaicin
Dietary Supplement: Piperine — Oral stimulation with natural TRPA1/V1 agonist
  Arms: Piperine
Dietary Supplement: Placebo — Oral stimulation with placebo solution
  Arms: Placebo

SUMMARY:
In recent years, the investigators have characterized the impairments in pharyngeal sensory function associated with swallowing disorders in older patients with oropharyngeal dysphagia (OD). The investigators have demonstrated the acute and sub-acute therapeutic effect of TRP agonists on mechanical and neural swallow responses in patients with OD. The present hypothesis is that 6-months treatment with TRPV1 (capsaicin) or TRPA1 (piperine) agonists will improve the biomechanics and neurophysiology of the swallow response without inducing desensitization. The aim of this study is to evaluate the effect on biomechanics assessed by videofluoroscopy (VFS), neurophysiology (pharyngeal evoked sensory potentials -pSEP- and motor evoked potentials -pMEP-), and clinical outcomes during a 6-month treatment with TRP agonists added to the alimentary bolus 3 times a day in older patients with OD. Design: 150 older patients (>70y) with OD will be included in a randomized clinical trial with three treatment arms, in which the effect of oral administration of 1) capsaicin 10µM (TRPV1 agonist), 2) piperine 150µM (TRPA1), and 3) placebo (Control), will be evaluated. Measurements: 1) VFS signs of swallowing safety and efficacy and timing of swallow response ; 2) Spontaneous swallowing frequency; 3) Latency, amplitude and cortical representation of pSEP and pMEP; 4) Concentration of substance P and CGRP in saliva, 5) Clinical outcomes (respiratory and nutritional complications). The results of this study will increase evidence for a new generation of pharmacological treatments for older patients with OD, moving from compensation to rehabilitation of the swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* ≥70 years
* With a positive Volume-Viscosity Swallow Test for oropharyngeal dysphagia
* Penetration-aspiration scale >1 in videofluoroscopy
* Able to follow the protocol and to give written informed consent.

Exclusion Criteria:

* Life expectancy < 3m or palliative care
* Allergy to iodinated contrast or to the components of the treatment solutions
* Cancer or active infection
* Implanted electronic device
* Epilepsy
* Metal in the head
* Participation in another clinical trial (previous month).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of oropharyngeal dysphagia | Pre treatment visit
  The severity of oropharyngeal dysphagia will be determined according the penetration-aspiration scale during the videofluoroscopy:
  1. Material does not enter the airway.
  2. Material enters the airway. Remains above vocal cords and is ejected from the airway.
  3. Material is above vocal cords and is not ejected from the airway.
  4. Material enters the airway, contacts vocal cords and is ejected from the airway.
  5. Material contacts the vocal cords and is not ejected from the airway.
  6. Material passes below the vocal cords and is ejected into larynx or out of the airway.
  7. Material passes below the vocal cords and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal cords and no effort is made to eject the material
Severity of oropharyngeal dysphagia | 1 month follow-up visit
  The severity of oropharyngeal dysphagia will be determined according the penetration-aspiration scale during the videofluoroscopy:
  1. Material does not enter the airway.
  2. Material enters the airway. Remains above vocal cords and is ejected from the airway.
  3. Material is above vocal cords and is not ejected from the airway.
  4. Material enters the airway, contacts vocal cords and is ejected from the airway.
  5. Material contacts the vocal cords and is not ejected from the airway.
  6. Material passes below the vocal cords and is ejected into larynx or out of the airway.
  7. Material passes below the vocal cords and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal cords and no effort is made to eject the material
Severity of oropharyngeal dysphagia | 3 month follow-up visit
  The severity of oropharyngeal dysphagia will be determined according the penetration-aspiration scale during the videofluoroscopy:
  1. Material does not enter the airway.
  2. Material enters the airway. Remains above vocal cords and is ejected from the airway.
  3. Material is above vocal cords and is not ejected from the airway.
  4. Material enters the airway, contacts vocal cords and is ejected from the airway.
  5. Material contacts the vocal cords and is not ejected from the airway.
  6. Material passes below the vocal cords and is ejected into larynx or out of the airway.
  7. Material passes below the vocal cords and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal cords and no effort is made to eject the material
Severity of oropharyngeal dysphagia | 6 month follow-up visit
  The severity of oropharyngeal dysphagia will be determined according the penetration-aspiration scale during the videofluoroscopy:
  1. Material does not enter the airway.
  2. Material enters the airway. Remains above vocal cords and is ejected from the airway.
  3. Material is above vocal cords and is not ejected from the airway.
  4. Material enters the airway, contacts vocal cords and is ejected from the airway.
  5. Material contacts the vocal cords and is not ejected from the airway.
  6. Material passes below the vocal cords and is ejected into larynx or out of the airway.
  7. Material passes below the vocal cords and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal cords and no effort is made to eject the material
Safety impairment signs | Pre treatment visit
  Prevalence of safety impairment signs (penetrations and/or aspirations) according to videofluoroscopic results
Safety impairment signs | 1 month follow-up visit
  Prevalence of safety impairment signs (penetrations and/or aspirations) according to videofluoroscopic results
Safety impairment signs | 3 month follow-up visit
  Prevalence of safety impairment signs (penetrations and/or aspirations) according to videofluoroscopic results
Safety impairment signs | 6 month follow-up visit
  Prevalence of safety impairment signs (penetrations and/or aspirations) according to videofluoroscopic results
Efficacy impairment signs | Pre treatment visit
  Prevalence of efficacy impairment signs (oral and pharyngeal residue) according to videofluoroscopic results
Efficacy impairment signs | 1 month follow-up visit
  Prevalence of efficacy impairment signs (oral and pharyngeal residue) according to videofluoroscopic results
Efficacy impairment signs | 3 month follow-up visit
  Prevalence of efficacy impairment signs (oral and pharyngeal residue) according to videofluoroscopic results
Efficacy impairment signs | 6 month follow-up visit
  Prevalence of efficacy impairment signs (oral and pharyngeal residue) according to videofluoroscopic results
Swallow biomechanics | Pre treatment visit
  Measurement of the timing of oropharyngeal swallow response during the videofluoroscopy:
  * Time to laryngeal vestibule closure
  * Time to upper esophageal sphincter opening
  * Time to laryngeal vestibule opening
Swallow biomechanics | 1 month follow-up visit
  Measurement of the timing of oropharyngeal swallow response during the videofluoroscopy:
  * Time to laryngeal vestibule closure
  * Time to upper esophageal sphincter opening
  * Time to laryngeal vestibule opening
Swallow biomechanics | 3 month follow-up visit
  Measurement of the timing of oropharyngeal swallow response during the videofluoroscopy:
  * Time to laryngeal vestibule closure
  * Time to upper esophageal sphincter opening
  * Time to laryngeal vestibule opening
Swallow biomechanics | 6 month follow-up visit
  Measurement of the timing of oropharyngeal swallow response during the videofluoroscopy:
  * Time to laryngeal vestibule closure
  * Time to upper esophageal sphincter opening
  * Time to laryngeal vestibule opening
Pharyngeal sensory evoked potential (pSEP) | Pre treatment visit
  pSEP will be recorded with a 32-electrode EEG recording cap (10/20 system) during a series of electrical stimuli applied to the pharynx with an intra-pharyngeal catheter.
Pharyngeal sensory evoked potential (pSEP) | 1 month follow-up visit
  pSEP will be recorded with a 32-electrode EEG recording cap (10/20 system) during a series of electrical stimuli applied to the pharynx with an intra-pharyngeal catheter.
Pharyngeal sensory evoked potential (pSEP) | 3 month follow-up visit
  pSEP will be recorded with a 32-electrode EEG recording cap (10/20 system) during a series of electrical stimuli applied to the pharynx with an intra-pharyngeal catheter.
Pharyngeal sensory evoked potential (pSEP) | 6 month follow-up visit
  pSEP will be recorded with a 32-electrode EEG recording cap (10/20 system) during a series of electrical stimuli applied to the pharynx with an intra-pharyngeal catheter.
Pharyngeal motor evoked potentials (pMEP) | Pre treatment visit
  pMEPs for both brain hemispheres will be recorded with an intra-pharyngeal catheter by applying 10 pulses of transcraneal magnetic stimulus to each hotspot (tenar and pharyngeal).
Pharyngeal motor evoked potentials (pMEP) | 1 month follow-up visit
  pMEPs for both brain hemispheres will be recorded with an intra-pharyngeal catheter by applying 10 pulses of transcraneal magnetic stimulus to each hotspot (tenar and pharyngeal).
Pharyngeal motor evoked potentials (pMEP) | 3 month follow-up visit
  pMEPs for both brain hemispheres will be recorded with an intra-pharyngeal catheter by applying 10 pulses of transcraneal magnetic stimulus to each hotspot (tenar and pharyngeal).
Pharyngeal motor evoked potentials (pMEP) | 6 month follow-up visit
  pMEPs for both brain hemispheres will be recorded with an intra-pharyngeal catheter by applying 10 pulses of transcraneal magnetic stimulus to each hotspot (tenar and pharyngeal).

SECONDARY OUTCOMES:
Spontaneous swallowing frequency (SSF) | Pre treatment visit and 1, 3 and 6 month follow-up visits
  SSF will be measured with surface neck electromyography and accelerometry for 10min to assess: the number of swallows per minute
Clinical outcomes: Hospital readmission rate | Pre treatment visit and 1, 3 and 6 month follow-up visits
  Hospital readmissions (readmissions/100 persons-year)
Clinical outcomes: Prevalence of lower respiratory tract infections | Pre treatment visit and 1, 3 and 6 month follow-up visits
  Lower respiratory tract infections (including pneumonia)
Clinical outcomes: Mortality | Pre treatment visit and 1, 3 and 6 month follow-up visits
  Mortality rate
Responders rate | 6 month follow-up visit
  Responders were defined as those patients who, after treatment, achieved safe swallow at a lower level of viscosity or, at the same viscosity level, improved at least one point in the penetration-aspiration scale.
Treatment palatability: Taste | 1, 3 and 6 month follow-up visits
  Facial scales on the palatability of the treatment will be performed from V2 to V4. Participants will be asked to respond to questions about the taste using the Face Likert scale: 1. Awful; 2. Not very good; 3. Okay; 4. Really good; 5. Fantastic.
Treatment palatability: Texture | 1, 3 and 6 month follow-up visits
  Facial scales on the palatability of the treatment will be performed from V2 to V4. Participants will be asked to respond to questions about the texture using the Face Likert scale: 1. Awful; 2. Not very good; 3. Okay; 4. Really good; 5. Fantastic.
Treatment palatability: Future Adherence | 1, 3 and 6 month follow-up visits
  Facial scales on the palatability of the treatment will be performed from V2 to V4. Participants will be asked to respond to questions about the possible future adherence to the treatment if prescribed using the Face Likert scale: 1. Awful; 2. Not very good; 3. Okay; 4. Really good; 5. Fantastic.
Salivary neuropeptides | 1, 3 and 6 month follow-up visits
  Saliva samples will be collected in all study visits using the Salivette® technique, by putting a swab under the tongue for 5 min. The concentration of salivary neuropeptides substance P (SP) and calcitonin gene-related peptide (CGRP) will be determined by using 2 specific commercial Enzyme-Linked ImmunoSorbent Assay (ELISA) kits
Treatment safety | From the inclusion to the study until the end of their participation (6 month)
  Adverse events occurring during the study will be monitored according to the guideline of categories described by the world health organization
Treatment compliance | Pre treatment visit and 1, 3 and 6 month follow-up visits
  A sample of urine will be collected at each study visit and the concentration of riboflavin (part of the composition of the product from the 3 groups) will be extrapolated with fluorescence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Mataró, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No